CLINICAL TRIAL: NCT06256302
Title: Transverses Abdominis Plane Block Versus Local Wound Infiltration for Postoperative Pain Management in Patients Undergoing Total Abdominal Hysterectomy
Brief Title: Transverses Abdominis Plane Block Versus Local Wound Infiltration in Total Abdominal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Muhammad Arif (Other)
Responsible Party: Sponsor-Investigator, Dr Muhammad Arif, Principal Investigator, Ziauddin University
Organization: Ziauddin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 7861023MAANE
Record Dates: First submitted 2024-02-01; First posted 2024-02-13 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Pain
Keywords: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transverses abdominis plane block (Experimental)
  Interventions: Procedure: Transverses Abdominis Plane Block
- Local wound infiltration (Active Comparator)
  Interventions: Procedure: Local wound infiltration

INTERVENTIONS:
Procedure: Transverses Abdominis Plane Block — Transverses abdominis plane block will be provided randomly using prospective double-blinding.
  Arms: Transverses abdominis plane block
Procedure: Local wound infiltration — Local wound infiltration will be provided randomly using prospective double-blinding.
  Arms: Local wound infiltration

SUMMARY:
To compare the transverses abdominis plane block outcome versus local wound infiltration for postoperative analgesia in patients undergoing total abdominal hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18 to 50 years
* Female
* ASA I & II
* Undergoing Abdominal Hysterectomy under General anaesthesia

Exclusion Criteria:

* Hepatic failure (assessed on clinical signs and symptoms, elevated liver enzymes and ultrasound findings showing loss of normal texture of liver) or renal failure (a GFR of 15 or less)
* Allergy or contraindication to study drugs on history
* Drug abuse or addiction
* Bleeding tendency

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Pain score | 24 hours of surgery.
  Pain score will be evaluated through Visual analogue scale (VAS) score of 0-10cms.

SECONDARY OUTCOMES:
Analgesia consumption | During 24 hours of surgery
  Patients will be given analgesics only on complain of pain of VAS score of 4 and above.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Arif, Principal Investigator — Ziauddin University
Locations (1):
- Muhammad Arif, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No